CLINICAL TRIAL: NCT00002181
Title: Open-Label Study of Cidofovir Gel for Acyclovir-Unresponsive Mucocutaneous Herpes Simplex Disease in Patients With AIDS.
Brief Title: Cidofovir as a Treatment for Herpes Simplex in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 218B; GS-96-307
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-11

CONDITIONS: Herpes Simplex; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Herpes Simplex; Acyclovir; Antiviral Agents; Gels; cidofovir
MeSH Terms: conditions — Herpes Simplex; HIV Infections; AIDS-Related Opportunistic Infections | interventions — Cidofovir

INTERVENTIONS:
Drug: Cidofovir

SUMMARY:
The purpose of this study is to see if cidofovir gel (Forvade) is safe and effective in treating herpes simplex in patients with AIDS who do not respond to acyclovir.

DETAILED DESCRIPTION:
Patients receive open-label treatment with cidofovir gel.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS diagnosis per CDC criteria.
* At least partially external mucocutaneous HSV infection confirmed by culture of current outbreak.
* Current HSV outbreak that is unresponsive to >= 10-day course of acyclovir at 1-4 gm/day po or 15 mg/kg/day IV or in vitro resistance of HSV isolate to acyclovir demonstrated within 60 days of study.
* Signed, informed consent from parent or legal guardian for patients less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

Evidence of cervical intraepithelial neoplasia class III (CIN III) on Pap smear (Pap smear required within 6 months of starting study drug).

Concurrent Medication:

Excluded:

Acyclovir, valacyclovir, famciclovir, ganciclovir, foscarnet, topical trifluride, cidofovir injection or other systemic or topical drugs with anti-herpes activity.

Required:

>= 10 day course acyclovir at 1-4 gm/day po or 15mg/kg/day IV (not required if there is confirmed in vitro resistance to acyclovir).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Mem Med Group Inc, Long Beach, California
  - AIDS Healthcare Foundation Labs, Los Angeles, California
  - Sharp Mission Park / Med Group, Oceanside, California
  - Park Ctr for Health / Keith Vrhel, San Diego, California
  - Potrero Hill Med Ctr, San Francisco, California
  - HIV Primary Care & Consult, Santa Rosa, California
  - Central Florida Research Initiative, Maitland, Florida
  - Braude Mermin Spivey MD PC, Atlanta, Georgia
  - Christie Clinic / Urbana Campus, Urbana, Illinois
  - Heywood Memorial Hosp, Gardner, Massachusetts
  - Gouverneur Hosp, New York, New York
  - Central Texas Med Foundation, Austin, Texas
  - Dr Nicholaos Bellos, Dallas, Texas
  - Dr Susan M Diamond, Dallas, Texas
  - ID Associates, Dallas, Texas